CLINICAL TRIAL: NCT00519012
Title: Prospective 24-week Study, Comparing Clinical Outcomes Between Switching Antidepressants and Maintaining the Same Antidepressant in Patients With Major Depressive Disorder Who do Not Show a 20% Reduction in Symptoms at Week 2
Brief Title: Benefits of Switching Antidepressants Following Early Nonresponse
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oizumi Hospital (Other)
Responsible Party: Shinichiro Nakajima, Keio university
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19760629
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Depression
Keywords: early nonresponse
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm-1 (Active Comparator): Sertraline to Paroxetine
  Interventions: Drug: Sertraline to Paroxetine
- 2 (Active Comparator): Paroxetine to Sertraline
  Interventions: Drug: Paroxetine to Sertraline

INTERVENTIONS:
Drug: Sertraline to Paroxetine — For subjects enrolled in this arm, sertraline will be initiated at 25mg, increased to 50mg on day 3, and maintained until day 14. If subjects show an early response (i.e. a 20% improvement in the MADRS total score from baseline) at week 2, sertraline will be continued and titrated at 50 - 100mg based on clinical judgment. On the other hand, if subjects fail to show an early response at week 2, they will be randomly divided into two groups. In one group, sertraline will be continued and titrated at 50 - 100mg, whereas in the other group sertraline will be switched to paroxetine. In this switching group, paroxetine will be started at 10mg on days 15 and 16, increased to 20mg on day 17, and further increased to 40mg by a weekly 10mg increase, while sertraline will be dosed at 25mg on day 15 and terminated on day 16.
  Arms: Arm-1
Drug: Paroxetine to Sertraline — Paroxetine will be initiated at 10mg, increased to 20mg on day 3, and maintained until day 14. If subjects show an early response (i.e. a 20% improvement in the MADRS total score from baseline) at week 2, paroxetine will be continued and titrated at 20 - 40mg based on clinical judgment. On the other hand, if subjects fail to show an early response at week 2, they will be randomly divided into two groups. In one group, paroxetine will be continued and titrated at 20 - 40mg, whereas in the other group paroxetine will be switched to sertraline. In this switching group, sertraline will be started at 25mg on days 15 and 16, increased to 50mg on day 17, and further increased to 100mg by a weekly 25mg increase, while paroxetine will be dosed at 10mg on day 15 and terminated on day 16.
  Arms: 2

SUMMARY:
Introduction and Purpose:

Most of the guidelines for the treatment of major depression recommend the use of antidepressants for 4 to 8 weeks. On the other hand, it has been recently reported that they start to show their antidepressant efficacy within a couple of weeks (1,2), contrary to the conventional theory. In addition, a good response (i.e. a 20% reduction in the Montgomery-Åsberg Depression Rating Scale [MADRS]) at week 2 is proposed to be a predictor of subsequent remission at week 6 (3,4), while nonresponse at week 2 could predict unfavourable outcome at week 8 (5). Furthermore, early worsening is suggested to be related to a low rate of remission at weeks 8 and 12(6).

DETAILED DESCRIPTION:
To the researchers' knowledge, there is no report to prospectively examine the benefits of switching antidepressants following early nonresponse. In this prospective 24-week study, the researchers will compare clinical outcomes between switching antidepressants and maintaining the same antidepressant in patients with major depressive disorder who do not show a 20% reduction in symptoms at week 2.

Materials and Methods: This open-label 24-week randomized controlled trial will be performed at psychiatric hospitals in Tokyo, Japan.

This study will be conducted with the approval of the Institutional Review Board of each participating hospital, and written informed consent will be obtained from all of the participants after providing a full explanation about the study.

In the short-term acute phase, sertraline will be initiated at 25 mg, increased to 50 mg on day 3, and maintained until day 14. If patients show an early response (i.e. ≧ 20% improvement in the MADRS total score from baseline), sertraline will be continued and titrated at 50 - 100 mg based on clinical judgment. On the other hand, if patients show no early response, they will be randomly divided into two groups. In one group, sertraline will be continued and titrated at 50 - 100 mg, whereas in the other group sertraline will be switched to paroxetine. Paroxetine will be started at 10 mg on days 15 and 16, increased to 20 mg on day 17, and further increased weekly by 10 mg from week 4 (i.e. day 22), while sertraline will be tapered by 25 mg each on days 15 and 16. In case patients are intolerant to adverse events, or they achieve remission (i.e. the MADRS total score ≦ 8), increasing the dose will be terminated. Lorazepam, lormetazepam, and mosapride will be allowed on a p.r.n. basis.

In the long-term follow-up phase after week 8, patients who achieve remission or response will be followed up and the same dose will be administered throughout. Assessments will include the MADRS, the clinical global impression scale (CGI), and the Quick Inventory of Depressive Symptomatology self-reported (QIDS-SR) (weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24). Adverse events will also be monitored on every visit.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients and outpatients who meet the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria of major depression disorder (MDD)
2. Have not taken antidepressants for the previous one month
3. Do not have emergent suicidal ideation defined as a score of 4 or less on suicidal thoughts item in the MADRS.

Exclusion Criteria

1. Unstable physical illness or clinically significant neurological disorder
2. Having emergent suicidal idea defined as a score of 5 or more on the suicidal thoughts item in the MADRS.
3. Having history of non-response or intolerance to paroxetine or sertraline.

This study will be conducted with the approval of the Institutional Review Board of each participating hospital, and written informed consent will be obtained from all of the participants after providing a full explanation of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-08; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The Montgomery-Asberg Depression Rating Scale | at weeks1, 2, 3, 4, 6, 8, 12, 16, 20, 24 and 48 - 52.

SECONDARY OUTCOMES:
The Clinical Global Impression 2. The Quick Inventory of Depressive Symptomatology self-reported | at weeks1, 2, 3, 4, 6, 8, 12, 16, 20, 24 and 48 - 52.

CONTACTS AND LOCATIONS:
Overall Officials: Shinichiro Nakajima, M.D., Study Chair — Oizumi Hospital
Locations (1):
- Oizumi Hospital, 6-9-1 Oizumigakuen-cho, Nerima-ku, Tokyo, Japan

REFERENCES:
- [Background] Papakostas GI, Perlis RH, Scalia MJ, Petersen TJ, Fava M. A meta-analysis of early sustained response rates between antidepressants and placebo for the treatment of major depressive disorder. J Clin Psychopharmacol. 2006 Feb;26(1):56-60. doi: 10.1097/01.jcp.0000195042.62724.76. PMID 16415707
- [Background] Taylor MJ, Freemantle N, Geddes JR, Bhagwagar Z. Early onset of selective serotonin reuptake inhibitor antidepressant action: systematic review and meta-analysis. Arch Gen Psychiatry. 2006 Nov;63(11):1217-23. doi: 10.1001/archpsyc.63.11.1217. PMID 17088502
- [Background] Katz MM, Tekell JL, Bowden CL, Brannan S, Houston JP, Berman N, Frazer A. Onset and early behavioral effects of pharmacologically different antidepressants and placebo in depression. Neuropsychopharmacology. 2004 Mar;29(3):566-79. doi: 10.1038/sj.npp.1300341. PMID 14627997
- [Background] Szegedi A, Muller MJ, Anghelescu I, Klawe C, Kohnen R, Benkert O. Early improvement under mirtazapine and paroxetine predicts later stable response and remission with high sensitivity in patients with major depression. J Clin Psychiatry. 2003 Apr;64(4):413-20. doi: 10.4088/jcp.v64n0410. PMID 12716243
- [Background] Nierenberg AA, McLean NE, Alpert JE, Worthington JJ, Rosenbaum JF, Fava M. Early nonresponse to fluoxetine as a predictor of poor 8-week outcome. Am J Psychiatry. 1995 Oct;152(10):1500-3. doi: 10.1176/ajp.152.10.1500. PMID 7573590
- [Background] Cusin C, Fava M, Amsterdam JD, Quitkin FM, Reimherr FW, Beasley CM Jr, Rosenbaum JF, Perlis RH. Early symptomatic worsening during treatment with fluoxetine in major depressive disorder: prevalence and implications. J Clin Psychiatry. 2007 Jan;68(1):52-7. doi: 10.4088/jcp.v68n0107. PMID 17284130